CLINICAL TRIAL: NCT04276129
Title: Early Healing of Oral Soft Tissues: a Clinical and Biomolecular Analysis. Part II - Effect of Local Chlorhexidine Administration in Gene Expression and Cellular Behaviour 24-hours After Injury
Brief Title: Early Healing of Oral Soft Tissues: a Clinical and Biomolecular Analysis. Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5315 Prot 1066/19
Record Dates: First submitted 2020-02-16; First posted 2020-02-19 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Wound Heal; Wound Surgical; Oral Soft Tissue Conditions; Chlorhexidine Adverse Reaction
Keywords: early wound healing; real-time polymerase chain reaction; gingiva; oral mucosa; palatal tissue; Chlorhexidine
MeSH Terms: conditions — Surgical Wound | interventions — Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post-surgical CHX mouth-rinses (treatment group - CHX) (Experimental): periodontal surgery + post-surgical CHX mouth-rinses + buccal attached gingival (G) biopsies 24 hr after surgical procedure
  Interventions: Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy; Other: post-surgical CHX mouth-rinses indication
- NO post-surgical mouth-rinses treatment (non treatment group - NT) (Other): periodontal surgery + buccal attached gingival (G) biopsies 24 hr after surgical procedure
  Interventions: Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy

INTERVENTIONS:
Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy — Periodontal surgery will be performed and 24 hr after the surgical procedure a 2mm punch biopsy will be harvested at the level of the buccal attache gingiva (G).
Other: post-surgical CHX mouth-rinses indication — CHX mouth-rinses (0.12%) will be indicated 2 times/day after the surgical procedure
  Arms: post-surgical CHX mouth-rinses (treatment group - CHX)

SUMMARY:
The purpose of the present study is to evaluate the influence of the post-surgical chlorhexidine indication in the gene expression profile and cellular behavior in the early wound healing process -24 hours after injury- of the oral soft tissues.

The main hypothesis is that the post-surgical use of chlorhexidine affects the gene expression and the celular behavior in the early wound healing process of the soft oral tissues.

DETAILED DESCRIPTION:
The bacterial infection control in the wound healing is a very important aspect to considerer. Local antiseptic administration after the surgical procedures has been used to control the bacterial contamination.

Chlorhexidine (CHX), widely used as antiseptic, especially as post-surgical indication, has a toxic effect both in vivo and in vitro and their influence on wound healing has been studied for a long time. One of the first animal studies, in 1980, concluded that intensive rinsing with high concentrations of chlorhexidine after oral surgical operations, could result in delay and disturbance of wound healing. Another more recent animal study concluded that CHX induces apoptosis or necrosis in the fibroblasts.

Mariotti and Rumpf, in 2016, carried out a studied incubating human gingival fibroblasts in CHX. The results have been suggested that chlorhexidine could induce a dose dependent reduction in cellular proliferation and that concentrations of chlorhexidine that have little effect on cellular proliferation can significantly reduce both collagen and non-collagen protein production of human gingival fibroblasts in vitro. Hence, the introduction of commercially available concentrations (0.12%) or diluted commercial concentrations (as low as 0.00009%) of chlorhexidine to surgical sites for short periods of time prior to wound closure can conceivably have serious toxic effects on gingival fibroblasts and may negatively affect wound healing.

All the previous mentioned studies permit understand that the CHX is not harmless to the oral tissues. However, its effect is not entirely clear and should be evaluated in depth taking into account that it is one of the most indicated antiseptics after surgery. Currently, there are no studies that evaluate if the post-surgical use of CHX affect the gene expression in the early wound healing.

ELIGIBILITY:
Inclusion Criteria:

* patients that required periodontal surgery;
* patients age between 30-60 years;
* patients with full mouth plaque score and full mouth bleeding score < 15%;
* patients with a good general healthy status;
* patients without any medicaments or drug consumption that can affect the healing process;
* non-smoking patients.

Exclusion Criteria:

* patients in pregnancy;
* patients in lactation period;
* patients with consumption of antibiotics or anti-inflammatory drugs in the previous six months;
* patients with systemic diseases.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Changes from baseline fold regulation wound healing related genes at 24 hours after post-surgical chlorhexidine use. | 24 hours after surgery (T24)
  Total RNA from biopsies or cell cultures was extracted using TRIzol reagent Quantitative real-time PCR (qRT-PCR) cDNA was generated and cDNA obtained were used for amplification of wound healing related genes using the appropriate TaqMan gene expression assay kits.

SECONDARY OUTCOMES:
Clinical evaluation of early wound healing | 24 hours after surgery (T24)
  Assessed with a clinical index (EHS- Early wound healing score). This score assessed clinical signs of re-epithelialization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Since complete wound epithelialization was the main outcome, the CSR score was weighted to be 60% of the total final score. Accordingly, a score of 0, 3, or 6 points was possible for the assessment of CSR, whereas scores of 0, 1, or 2 points were possible for CSH and CSI. Higher values indicated better healing. Accordingly, the score for ideal early wound healing was 10.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD,DDS,MS, Study Director — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillofacial Sciences. Section of Periodontics.Sapienza, University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eming SA, Martin P, Tomic-Canic M. Wound repair and regeneration: mechanisms, signaling, and translation. Sci Transl Med. 2014 Dec 3;6(265):265sr6. doi: 10.1126/scitranslmed.3009337. PMID 25473038
- [Result] Warburton G, Nares S, Angelov N, Brahim JS, Dionne RA, Wahl SM. Transcriptional events in a clinical model of oral mucosal tissue injury and repair. Wound Repair Regen. 2005 Jan-Feb;13(1):19-26. doi: 10.1111/j.1067-1927.2005.130104.x. PMID 15659033
- [Result] Mak K, Manji A, Gallant-Behm C, Wiebe C, Hart DA, Larjava H, Hakkinen L. Scarless healing of oral mucosa is characterized by faster resolution of inflammation and control of myofibroblast action compared to skin wounds in the red Duroc pig model. J Dermatol Sci. 2009 Dec;56(3):168-80. doi: 10.1016/j.jdermsci.2009.09.005. Epub 2009 Oct 24. PMID 19854029
- [Result] Iglesias-Bartolome R, Uchiyama A, Molinolo AA, Abusleme L, Brooks SR, Callejas-Valera JL, Edwards D, Doci C, Asselin-Labat ML, Onaitis MW, Moutsopoulos NM, Gutkind JS, Morasso MI. Transcriptional signature primes human oral mucosa for rapid wound healing. Sci Transl Med. 2018 Jul 25;10(451):eaap8798. doi: 10.1126/scitranslmed.aap8798. PMID 30045979
- [Result] Wang Y, Tatakis DN. Human gingiva transcriptome during wound healing. J Clin Periodontol. 2017 Apr;44(4):394-402. doi: 10.1111/jcpe.12669. Epub 2017 Feb 11. PMID 28005267
- [Result] Vescarelli E, Pilloni A, Dominici F, Pontecorvi P, Angeloni A, Polimeni A, Ceccarelli S, Marchese C. Autophagy activation is required for myofibroblast differentiation during healing of oral mucosa. J Clin Periodontol. 2017 Oct;44(10):1039-1050. doi: 10.1111/jcpe.12767. Epub 2017 Aug 25. PMID 28646601
- [Result] Marini L, Rojas MA, Sahrmann P, Aghazada R, Pilloni A. Early Wound Healing Score: a system to evaluate the early healing of periodontal soft tissue wounds. J Periodontal Implant Sci. 2018 Oct 24;48(5):274-283. doi: 10.5051/jpis.2018.48.5.274. eCollection 2018 Oct. PMID 30405935
- [Result] Bassetti C, Kallenberger A. Influence of chlorhexidine rinsing on the healing of oral mucosa and osseous lesions. J Clin Periodontol. 1980 Dec;7(6):443-56. doi: 10.1111/j.1600-051x.1980.tb02151.x. PMID 6938525
- [Result] Faria G, Cardoso CR, Larson RE, Silva JS, Rossi MA. Chlorhexidine-induced apoptosis or necrosis in L929 fibroblasts: A role for endoplasmic reticulum stress. Toxicol Appl Pharmacol. 2009 Jan 15;234(2):256-65. doi: 10.1016/j.taap.2008.10.012. Epub 2008 Nov 6. PMID 19027770
- [Result] Mariotti AJ, Rumpf DA. Chlorhexidine-induced changes to human gingival fibroblast collagen and non-collagen protein production. J Periodontol. 1999 Dec;70(12):1443-8. doi: 10.1902/jop.1999.70.12.1443. PMID 10632519